CLINICAL TRIAL: NCT02445781
Title: Mechanisms of Hypoglycemia Associated Autonomic Dysfunction, Differing Levels of Hypoglycemia
Brief Title: Differing Levels of Hypoglycemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Chairman of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 00064405
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 90 mg/dl glucose clamp (Experimental): Glucose clamp intervention of 90 mg/dl maintained for 90 minutes.
  Interventions: Device: Glucose clamp
- 70 mg/dl glucose clamp (Experimental): Glucose clamp intervention of 70 mg/dl maintained for 90 minutes.
  Interventions: Device: Glucose clamp
- 60 mg/dl glucose clamp (Experimental): Glucose clamp intervention of 60 mg/dl maintained for 90 minutes.
  Interventions: Device: Glucose clamp
- 50 mg/dl glucose clamp (Experimental): Glucose clamp intervention of 50 mg/dl maintained for 90 minutes.
  Interventions: Device: Glucose clamp

INTERVENTIONS:
Device: Glucose clamp — Different levels of hypoglycemia

SUMMARY:
Hypoglycemia can produce a spectrum of pro-inflammatory and pro-atherothrombotic changes. To date no studies appear to have investigated the effects of differing levels of hypoglycemia on the vasculature and pro-atherothrombotic balance during hypoglycemia in healthy man. The specific aim of our study will be to determine the effects of differing levels of hypoglycemia on in-vivo vascular biologic mechanisms in a healthy population.

DETAILED DESCRIPTION:
Recent large randomized multicenter trials have investigated the effects of lowering blood glucose levels towards normal in both inpatient and ambulatory care/community settings. All studies have reported increasing prevalence and incidence of hypoglycemia as glucose levels approach normal. In fact, the occurrence of hypoglycemia was so problematic that some hospital based studies were halted and the target recommendations for glucose levels in critically unwell patients have been increased. Similarly three recent large glucose control and complications trials in type 2 diabetes mellitus (DM) have reported significantly high rates of hypoglycemia in intensively treated type 2 DM individuals. In two of these studies (VADT, ADVANCE) there was a highly significant association between severe hypoglycemia (glucose low enough to cause neurologic impairment) and serious cardiac events and increased death. Furthermore, in two studies performed in the USA (VADT, ACCORD), severe hypoglycemia occurring in the standard/conventionally treated group produced even more serious adverse cardiac effects as compared to the intensively treated group. The in-vivo mechanism(s) responsible for the above findings could not be identified from the above studies. Surprisingly there is very limited data available regarding the effects of hypoglycemia on in-vivo vascular biology. Previously, in vitro work has determined that epinephrine, norepinephrine, growth hormone, glucagon, and corticosteroids (all counterregulatory hormones) can have vascular biologic effects (platelet aggregation, fibrinolytic balance, increases in pro-inflammatory markers and changes in endothelial function). Three recent studies from my own and other laboratories performed in healthy volunteers and type 1 DM have demonstrated that hypoglycemia can produce a spectrum of pro-inflammatory and pro-atherothrombotic changes. Novel preliminary data from my lab has also demonstrated that hypoglycemia can impair endothelial function, reduce fibrinolytic balance (increase plasminogen activator inhibitor-1) and produce pro-atherothrombotic (increase platelet aggregation, thrombin anti-thrombin complexes, vascular adhesion molecules) changes in type 2 DM. Additionally, preliminary data presented below will demonstrate that a 90 minute episode of hypoglycemia (50 mg/dl) produces similar pro-atherothrombotic changes as compared to 4 hours of hyperglycemia (200 mg/dl). However, as investigators are just beginning to realize the effects of hypoglycemia on vascular biology, there remain many unanswered questions. For example, in the vulnerable type 2 DM population what is the dose response of different levels of hypoglycemia with attendant ANS activation on endothelial function and atherothrombotic balance? How does level of glycemic control affect ANS and vascular biologic responses to hypoglycemia in type 2 DM? Proposed studies in this protocol will provide novel information answering the clinically important question regarding the effects of mild to moderate hypoglycemia on vascular biologic mechanisms in a healthy population.

ELIGIBILITY:
Inclusion Criteria:

• Body mass index >21kg · m-2

Exclusion Criteria:

* Pregnant women
* Subjects unwilling or unable to comply with approved contraception measures
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Subjects with a history of severe, uncontrolled hypertension, heart disease, cerebrovascular incidents
* Current tobacco use
* Subjects with any known allergies to any of the study medications being used

Physical Exam Exclusion Criteria

* Uncontrolled severe hypertension (i.e., blood pressure greater than 160/100)
* Clinically significant cardiac abnormalities (e.g. heart failure, arrhythmia)
* Pneumonia treatment or hospitalization within 2 weeks prior to enrollment (study visit)
* Hepatic failure / jaundice
* Renal failure
* Cerebrovascular accident occurrence or hospitalization within 4 weeks prior to enrollment
* Fever greater than 38.0 degrees C

Screening Laboratory Tests Exclusion Criteria

* Hematocrit lower than 32 %
* White blood cell (WBC) count lower than 3 thou/ul or greater than 14 thou/ul
* Liver function tests: serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) greater than twice upper limit of normal range
* Alkaline phosphatase greater than 150U/L
* Total bilirubin (TBil) greater than 2 mg/dl
* Estimated glomerular filtration rate (eGFR) less than 60 mL/min/1.73 m2
* Positive human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Any abnormal cardiac response during multi-stage exercise test (if over 40 years of age)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-07; Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Flow mediated vasodilation of brachial artery measurements (mean maximum % change) | 120 minutes (pre) clamp and 240 minutes (post) clamp
  baseline (pre) measurements compared to end of clamp (post) measurements

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States